CLINICAL TRIAL: NCT04260698
Title: An Open Label Expanded Access Study of Omidubicel, for Allogeneic Transplantation in Patients With Hematological Malignancies
Brief Title: Expanded Access of Omidubicel, for Allogeneic Transplantation in Patients With Hematological Malignancies
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gamida Cell ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GC P#07.01.020
Record Dates: First submitted 2020-02-05; First posted 2020-02-07 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Hematological Malignancies
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- omidubicel (Experimental): Omidubicel is a cryopreserved stem/progenitor cell based product comprised of:
  1. Ex vivo expanded, umbilical cord blood-derived hematopoietic CD34+ progenitor cells (cultured fraction (CF))
  2. the non-cultured cell fraction of the same Cord Blood Unit (CBU) (Non-cultured Fraction (NF)) consisting of mature myeloid and lymphoid cells.
  Both fractions, i.e. CF and NF, will be kept frozen until they are thawed and infused on the day of transplantation.
  Interventions: Biological: omidubicel

INTERVENTIONS:
Biological: omidubicel — hematopoietic stem cell transplant
  Other Names: NiCord

SUMMARY:
Omidubicel is an investigational therapy for patients with high-risk hematologic malignancies.

DETAILED DESCRIPTION:
Successful blood and marrow transplantation (BMT) requires the infusion of a sufficient number of hematopoietic stem/progenitor cells (HSPCs), capable of both homing to the bone marrow and regenerating a full array of hematopoietic cell lineages with early and late repopulating ability in a timely fashion.

Omidubicel is a stem/progenitor cell-based product composed of ex vivo expanded allogeneic cells from one entire unit of umbilical cord blood. Omidubicel utilizes the small molecule nicotinamide (NAM), as an epigenetic approach to inhibit differentiation and to increase the migration, bone marrow (BM) homing and engraftment efficiency of hematopoietic progenitor cells (HPC) expanded in ex vivo cultures.

The overall study objectives are to provide access to omidubicel for transplantation in patients with hematological malignancies and to collect additional safety and efficacy data.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be at least 12 years of age
* Applicable disease criteria
* Patients must have one or two partially HLA-matched CBUs
* Back-up stem cell source
* Sufficient physiological reserves
* Females of childbearing potential agree to use appropriate method of contraception
* Signed written informed consent

Exclusion Criteria:

* Extensive bone marrow fibrosis
* Donor specific anti-HLA antibodies
* Pregnancy
* Medically unsuitable for transplant

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-07-08 (Actual); Primary Completion 2025-05-08 (Actual); Study Completion 2025-05-08 (Actual)

PRIMARY OUTCOMES:
To assess the time from transplant to neutrophil engraftment | by day 42 post-transplant inclusive

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Horwitz, MD, Principal Investigator — Duke University
Locations (6):
- United States (6):
  - UCLA, Los Angeles, California
  - Stanford University Cancer Institute, Palo Alto, California
  - Loyola University, Cardinal Bernardin Cancer Center, Maywood, Illinois
  - University of Minnesota Masonic Cancer Center, Minneapolis, Minnesota
  - Duke University Medical Center, Durham, North Carolina
  - Oregon Health & Science University, Portland, Oregon

IPD SHARING:
Plan to Share IPD: No